CLINICAL TRIAL: NCT03703479
Title: The Effect of Advanced Platelet Rich Fibrin in Alveolar Defect After Removal of Bilateral Mandibular Third Molar
Brief Title: Effect of A-PRF After Removal of Wisdom Teeth
Acronym: A-PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, talal zahid, Assistant professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 085-10-17
Record Dates: First submitted 2018-10-08; First posted 2018-10-12 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Wound Heal

STUDY DESIGN:
Intervention Model Description: spilt mouth design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-PRF group (Experimental): Socket site that will receive A-PRF clot
  Interventions: Other: autologous blood clot made from the patient own clot without any additive
- control (No Intervention): socket site that will not receive any intervention

INTERVENTIONS:
Other: autologous blood clot made from the patient own clot without any additive — advanced Platelet-rich fibrin clot is made from venous blood withdrawn from the patient
  Arms: A-PRF group

SUMMARY:
To evaluate the healing effect of advanced platelet-rich fibrin (blood clot charged with growth factors) taken from the patient own blood on the extraction site.

DETAILED DESCRIPTION:
This is a randomized double-blind clinical study. A preoperative and radiographic evaluation will be done in order to select the patients.

Inclusion criteria are healthy patients above 18 years old with vertical or mesioangular bilateral impacted mandibular third molars. Exclusion criteria are missing second molars or indicated for extraction (un-restorable and remaining roots), patients under immunosuppressant and patients with acute infection. Those who fail to attend for follow-up appointments will be excluded.

The probing depth (PD) and clinical attachment level (CAL) distal to the second molar will be measured before each procedure. All patients will undergo bilateral removal of 3rd molar in a single appointment. Envelope flap with distal extension and a full-thickness mucoperiosteal flap will be utilized and the teeth will be removed with elevators. Bone removal will be utilized if needed.

Following the extraction, venous blood will be withdrawn to fill 2 tubes of 10mL each (sterile vacuum plain tube for A-PRF™ +). The blood tubes will be spun in the centrifugation machine for 13 minutes at 1300 rpm then it is pressed in PRF Box to form PRF clots which will be placed in one the extraction socket while the other socket will not receive a PRF (control).Randomization will be done using a coin toss.

Both extraction cavities will be closed using 3-4 interrupted sutures using 3.0 chromic gut sutures.

Postoperatively, all patients will be treated with oral antibiotic amoxicillin 500 mg and non-steroidal anti-inflammatory medications ibuprofen 600mg in case. also, all patients will be instructed to rinse with 0.2 % Chlorhexidine mouthwash for seven days postoperative.

On the 7th,15th and 90th days, patients will be asked about pain using visual analog scale (VAS) and whether they have any concern related to extraction socket statuses like halitosis, empty socket, open socket, dehiscence, and infection signs including swelling, pus, or fever.

They will also undergo a clinical examination at this visit and the consecutive visits. The following measures will be assessed during each clinical examination: the presence of a pocket distal to the adjacent second molar measuring the pocket depth and clinical attachment level and any signs of infection.

Data will be analyzed using statistical software. Analysis of multivariate regression will be used. The healing status will be compared between the graft site and the control site. Results will be interpreted to be statistically significant if they have a P-value of less than 0.05

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients above 18 years old with mirror image vertical or mesioangular bilateral impacted mandibular third molars

Exclusion Criteria:

* Missing second molars or indicated for extraction (un-restorable and remaining roots).
* Patients under immunosuppressant and patients with acute infection.
* Patients who fail to attend for follow-up appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-03-24 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Loss (CAL) (also called Periodontal Attachment Loss) | At baseline and at follow-up 4 weeks and 12 weeks after extraction
  Periodontal healing is evaluated based on changes in clinical attachment loss (mm)

SECONDARY OUTCOMES:
Pain reported by the patient according to the visual analogue scale (VAS) | 7 days after the extraction
  Pain reported by the patient according to the visual analogue scale (VAS) will be evaluated at first follow-up visit, the patient will score the pain suffered at each site on 0-10 scale where 0 = no pain and 10 = sever pain

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdul Aziz University, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zahid TM, Nadershah M. Effect of Advanced Platelet-rich Fibrin on Wound Healing after Third Molar Extraction: A Split-mouth Randomized Double-blind Study. J Contemp Dent Pract. 2019 Oct 1;20(10):1164-1170. PMID 31883251